CLINICAL TRIAL: NCT04805125
Title: Randomised Controlled Trials to Assess Approved SARS-CoV-2 Vaccines in Immunocompromised Patients: A Master Protocol for the Set-up of a Swiss Cohorts Based Trial Platform
Brief Title: Immunocompromised Swiss Cohorts Based Trial Platform
Acronym: COVERALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-000593; me20Bucher
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Immunocompromised Patients
Keywords: Covid-19 infection; SARS-CoV-2-specific antibodies; Sars-CoV-2 vaccine; vector based messenger ribonucleic acid (mRNA) vaccines; SARS-CoV-2 infection; Swiss HIV Cohort Study [SHCS]; Swiss Transplant Cohort Study [STCS]; BNT162b2; mRNA-1273; bivalent SARS-CoV-2 vaccine; mRNA-1273.214
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Cohort embedded platform with a first sub-study pilot trial of two arms comparing licensed vaccines against SARS-CoV-2. The platform design allows to expand the pilot trial into a larger trial by sub-protocols to add or drop vaccine arms or to add further sub-protocols for re-randomization of patients with no immune response to a vaccine booster or new vaccines A parallel two-arm open-label randomized controlled exploratory pilot trial comparing the first in Switzerland approved SARS-CoV-2 vaccines (based on a trial platform that is integrated into the ongoing routine prospective data collection of two national cohorts, the SHCS and STCS). Within substudy-2 and substudy-3 observational studies were added to the platform trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderna mRNA COVID-19 vaccine (Active Comparator): The Moderna COVID-19 Vaccine, mRNA-1273 (100 μg) is administered intramuscularly as a series of two doses (0.5 mL each), given 28 days apart.
  ARM CLOSED
  Interventions: Biological: Moderna COVID-19 Vaccine, mRNA-1273 (100 μg)
- Comirnaty® (Pfizer / BioNTech) mRNA COVID-19 vaccine (Active Comparator): Active:
  The comparator product is the first licensed vaccine against SARS-CoV-2 in Switzerland.
  Pfizer-BioNTech COVID-19 Vaccine, BNT162b2 (30 µg) Comirnaty®, is administered intramuscularly (IM) as a series of two 30 µg doses of the diluted vaccine solution (0.3 mL each) according to the following schedule: a single dose followed by a second dose 21 days later.
  ARM CLOSED
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine BNT162b2 (30 µg)( Comirnaty®)

INTERVENTIONS:
Biological: Moderna COVID-19 Vaccine, mRNA-1273 (100 μg) — intramuscular injection, proposed as a series of two doses (0.5 mL each), dosing is 100 microgram on day 0 and day 28
  Arms: Moderna mRNA COVID-19 vaccine
Biological: Pfizer-BioNTech COVID-19 Vaccine BNT162b2 (30 µg)( Comirnaty®) — intramuscular injection, proposed dosing is 30 microgram of the diluted vaccine solution (0.3 mL each) on day 0 and day 21
  Arms: Comirnaty® (Pfizer / BioNTech) mRNA COVID-19 vaccine

SUMMARY:
This study is to set up a flexible trial platform using two existing national cohorts of immunocompromised patients (i.e. Swiss HIV Cohort Study [SHCS] and Swiss Transplant Cohort Study [STCS]) to assess the comparative effectiveness and safety of approved SARS-CoV-2 vaccines in immunocompromised patients.

This platform will be tested in the frame of an exploratory pilot trial and a framework will be set up to conduct a larger, flexible, randomized controlled trial (RCT) to test approved SARS-CoV-2 vaccines to prevent SARS-CoV-2 infections.

The first sub-protocol for a pilot trial is to investigate the operability of a platform trial that is nested into two existing cohort studies and compare immune response, safety and clinical efficacy of the first two mRNA vaccines (Comirnaty® by Pfizer / BioNTech and COVID-19 mRNA Vaccine Moderna®, by Moderna) in immune compromised patients in the Swiss HIV and Swiss Transplant Cohort studies.

The second sub-protocol (observational study) is to collect a blood sample before the third vaccination and 8 weeks after vaccination to analyze an additional benefit of a third SARS-CoV-2 vaccine in these immunocompromised patients.

In the third sub-protocol (substudy-3; observational) we will recruit patients who have received m-RNA-1273.214 by Moderna in the frame of clinical routine. We will start a second arm of our observational study as soon as another bivalent mRNA vaccine (from Pfizer-BioNTech) has been approved by Swissmedic. We aim to compare the immunologic response and safety of the bivalent mRNA-1273.214 vaccine from Moderna among immunocompromised persons (persons living with HIV or kidney or lung transplant recipients) to the immunologic response of immunocompromised persons who received the bivalent mRNA vaccine from Pfizer-BioNTech.

DETAILED DESCRIPTION:
The aim of this study is to set up a flexible trial platform using two existing national cohorts of immunocompromised patients (i.e. Swiss HIV Cohort Study [SHCS] and Swiss Transplant Cohort Study [STCS]) to assess the comparative effectiveness and safety of approved SARS-CoV-2 vaccines in immunocompromised patients. Nesting this trial into cohorts with highly standardized data collection allows for a rapid, efficient and cost-saving trial conduct.

This platform will be tested in the frame of a pilot trial and a framework will be set up to conduct a larger, flexible, randomized controlled trial (RCT) to test approved SARS-CoV-2 vaccines to prevent SARS-CoV-2 infections.

The pilot study will primarily assess the functionality of the trial platform and early immunogenicity, efficacy and safety data. At a later stage, the platform might also be used to enlarge the pilot trial or to develop sub-protocols to deal with patients with no or insufficient immune response to Sars-CoV-2 vaccines.

Since January 12, 2021 two mRNA vaccines against Sars-CoV-2 by Pfizer / BioNTech (Comirnaty®) and COVID-19 mRNA Vaccine Moderna® by Moderna have been licensed in Switzerland and roll-out of vaccines has started

The first sub-protocol for a pilot trial is to investigate the operability of a platform trial that is nested into two existing cohort studies and compare immune response, safety and clinical efficacy of the first two mRNA vaccines (Comirnaty® by Pfizer / BioNTech and COVID-19 mRNA Vaccine Moderna®, by Moderna) in immune compromised patients in the Swiss HIV and Swiss Transplant Cohort studies.

In Switzerland, since October 2021 severely immunodeficient persons ≥ 12 years of age who have received two doses of an mRNA vaccine should receive a third dose of Comirnaty® or Spikevax® as part of the basic immunization, regardless of any antibody titer. Among all other immunocompromised patients a booster vaccination with an mRNA vaccine is recommended. These vaccines will be administered to patients from the SHCS and the STCS in the frame of clinical routine.

This second sub-protocol (observational study) is to collect a blood sample before the third vaccination and 8 weeks after vaccination to analyze an additional benefit of a third SARS-CoV-2 vaccine in these immunocompromised patients.

In the third sub-protocol (substudy-3; observational) we will recruit patients who have received m-RNA-1273.214 by Moderna in the frame of clinical routine. We will start a second arm of our observational study as soon as another bivalent mRNA vaccine (from Pfizer-BioNTech) has been approved by Swissmedic. We aim to compare the immunologic response and safety of the bivalent mRNA-1273.214 vaccine from Moderna (n=160) among immunocompromised persons (persons living with HIV or kidney or lung transplant recipients) to the immunologic response of immunocompromised persons who received the bivalent mRNA vaccine from Pfizer-BioNTech (n=80). Patients will be asked to provide blood sample at baseline (before receiving bivalent mRNA SARS-CoV-2 vaccine) and 4 weeks, 8 weeks, and 6 months after vaccination (see details in original study protocol below).

ELIGIBILITY:
Inclusion criteria:

* All patients registered with informed consent from participating cohorts aged ≥18 years
* Additional consent for participation in the specific sub-protocol trial

Inclusion criteria for pilot trial:

* All patients with either a chronic HIV infection or recipients of solid organs registered with informed consent from the SHCS and STCS cohorts aged ≥18 years
* Patients with solid organ transplantation of lungs or kidneys at least one month post-transplantation with a prednisone dose of 20mg or less.
* Covid-19 vaccination recommended by treating physician

Inclusion criteria for 2. sub protocol (observational study):

* Third covid-19 vaccination recommended by treating physician and administered in the frame of clinical routine

Inclusion criteria for 3. substudy.

- Patients receiving a new bivalent (Wuhan/Omicron BA.1) mRNA SARS-CoV-2 vaccine in the frame of clinical routine, according to the treating physician

Exclusion criteria:

* Acute symptomatic SARS-CoV-2 infection, influenza or other acute respiratory tract infection
* Known allergy or contra-indications for vaccines or any vaccine components
* Any emergency condition requiring immediate hospitalization for any condition
* Patients with previous PCR documented SARS-CoV-2 infection and, or documented antibodies less than 3 months prior to screening visit (day 0)

Exclusion criteria for pilot trial:

* Pregnancy
* Acute symptomatic SARS-CoV-2 infection, influenza or other acute respiratory tract infection
* Known allergy or contra-indications for vaccines or any vaccine components
* Any emergency condition requiring immediate hospitalization for any condition
* Patients with previous PCR documented SARS-CoV-2 infection and, or documented antibodies less than 3 months prior to randomisation
* Patients with solid organ transplantation (lung or kidney) with the following conditions:

  1. Solid organ transplant recipients less than one month post-transplantation
  2. Solid organ transplant recipients with the use of T-cell/B-cell depleting agents in the last 3 months (i. e induction treatment in standard risk or high-risk immunological situation or rejection treatment).
  3. Solid organ transplant recipients with the need of pulse corticosteroids (>100mg prednisone or equivalent) in the last 1 month or who have received ATG or rituximab in the last 6 months
  4. Solid organ transplant recipients with the need of any kind of chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
immunological outcome: change in pan-Ig antibody response (pan-Ig anti-S1-RBD) | at baseline (day of vaccination) and three months after vaccination
  A commercial immunoassay Elecsys® Anti-SARS-CoV-2 S for the in vitro quantitative determination of antibodies to the SARS-CoV-2 spike (S) protein receptor binding domain (RBD) in human serum and plasma is used. This assay detects pan-Ig antibody response (pan-Ig anti-S1-RBD) and allows for a quantitative assessment of the serological response of the participants.
immunological outcome: change in anti-Nucleocapsid (N) response | at baseline (day of vaccination) and three months after vaccination
  Qualitative measurement of anti-Nucleocapsid (N) responses with Elecsys® Anti-SARS-CoV-2 N assay
immunological outcome: change in SARS-CoV-2-binding antibodies | at baseline (day of vaccination) and three months after vaccination
  SARS-CoV-2-binding antibody responses of the participants are assessed by analyzing the IgM, IgA and IgG responses to a wider range of SARS-CoV-2 proteins (S1, S2, RBD and N) using an in-house method (ABCORA). The ABCORA test allows a parallel assessment of IgG, IgM and IgA reactivity.
Number of participants with newly polymerase chain reaction (PCR)-confirmed asymptomatic COVID-19 infection | at any time point in within 48 weeks following randomisation (day of vaccination)
  Number of participants with newly PCR-confirmed asymptomatic COVID-19 infection (identified by the presence of anti-SARS-CoV-2 nucleocapsid antibodies or Sars-Cov-2 PCR or rapid antigen test) and no related symptoms [(i.e. fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose nausea or vomiting, and diarrhea])
Number of participants with newly PCR-confirmed symptomatic COVID-19 infection | at any time point in within 48 weeks following randomisation (day of vaccination)
  Number of participants with newly PCR-confirmed symptomatic COVID-19 infection with at least one of the following symptoms (i.e. fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose nausea or vomiting, and diarrhea
Number of participants with severe COVID-19 infection | at any time point in within 48 weeks following randomisation (day of vaccination)
  Number of participants with severe COVID-19 infection with respiratory failure, evidence of shock (as diagnosed by a treating physician), clinically significant acute renal, hepatic, or neurologic dysfunction; admission to an intensive care unit; or death
Clinical Outcome: COVID-19 burden of diseases (BOD) | within 48 weeks following randomisation (day of vaccination)
  COVID-19 burden of diseases (BOD), a composite, will be scored as by using 0 for no COVID-19, 1 for non-severe COVID-19, and 2 for severe COVID-19.
Duration of RCT set up (specific endpoint related to trial conduct feasibility) | one time assessment at baseline (from deciding which interventions will be tested until the first patient is randomised)
  Duration of RCT set up (i.e. time from deciding which interventions will be tested until the first patient is randomised).
Time of patient recruitment from activation of first study site until 40 patients are randomised | one time assessment after approx. 3 months (from activation of first study site until 40 patients are randomised)
  Time of patient recruitment from activation of first study site until 40 patients are randomised
Time of patient recruitment from activation of first study site until 380 patients are randomised | one time assessment after approx. 3 months (from activation of first study site until 380 patients are randomised)
  Time of patient recruitment from activation of first study site until 380 patients are randomised
Patient consent rate | approx. 3 months
  Patient consent rate (i.e. proportion of patients giving informed consent out of approached eligible patients)
Proportion of missing data for all baseline variables from routinely collected cohort data | one time assessment at baseline
  Proportion of missing data for all baseline variables from routinely collected cohort data
Proportion of missing data for all clinical outcomes | one time assessment after approx. 3 months
  Proportion of missing data for all clinical outcomes from routinely collected cohort data and outcome data that is collected in the trial platform
SARS-CoV-2-specific antibodies | three months after vaccination
  SARS-CoV-2-specific antibodies (using a pan-IgG antibody assay against the receptor binding domain (RBD) against the nP and spike 1 subunits)
SARS-CoV-2-specific titers | three months after vaccination
  SARS-CoV-2-specific titers (using an in-house assay developed by the Institute of Medical Virology, University of Zurich which can detect multiple viral epitopes)
The proportion of patients with a positive antibody response to SARS-CoV-2 spike (S1) protein receptor binding domain in human serum or plasma assessed in the observational second sub- protocol | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  The proportion of patients with a positive antibody response to SARS-CoV-2 spike (S1) protein receptor binding domain in human serum or plasma assessed or plasma assessed in the observational second sub- protocol by the commercial immunoassay Elecsys Anti-SARS-CoV-2 S (Elecsys S) from Roche Diagnostics. An antibody response will be considered as positive using the threshold ≥ 100 units/ml, predicting a protective immune response.

SECONDARY OUTCOMES:
The proportion of patients with a positive antibody response using SARS-CoV-2 spike (S1) Elecsys S by Roche in the observational second sub- protocol, using a threshold of ≥0.8 units/ml as defined by the manufacturer | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  The proportion of patients with a positive antibody response using SARS-CoV-2 spike (S1) Elecsys S by Roche in the observational second sub- protocol, using a threshold of ≥0.8 units/ml as defined by the manufacturer
The proportion of patients with a positive antibody response using antibody response using the Antibody CORonavirus Assay (ABCORA) 2 in the observational second sub- protocol | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  The proportion of patients with a positive antibody response using antibody response using the Antibody CORonavirus Assay (ABCORA) 2 in the observational second sub- protocol that assesses seropositivity by measuring specific IgG, IgA and IgM responses to SARS-CoV-2 receptor binding domains, S1, S2 and N16
The proportion of patients with neutralizing neutralization activity against the vaccine strain Wuhan-Hu-1 in the observational second sub- protocol | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  The proportion of patients with neutralizing neutralization activity against the vaccine strain Wuhan-Hu-1 in sera in the observational second sub- protocol defined as having an ABCORA sum S1 (sum of S1 signal over cut-off values of IgG, IgA, IgM) above the threshold of 17.
Immune response (pan-Ig antibodies against the receptor binding domain (RBD) in the S1 subunit of the spike protein (pan-Ig anti-S1-RBD) of SARS-CoV-2 in the observational second sub- protocol | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  Immune response (pan-Ig antibodies against the receptor binding domain (RBD) in the S1 subunit of the spike protein (pan-Ig anti-S1-RBD) of SARS-CoV-2 in the observational second sub- protocol
Mean immune response of IgM, IgA and IgG to the subunit S1 using ABCORA in the observational second sub- protocol | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  Mean immune response of IgM, IgA and IgG to the subunit S1 using ABCORA in the observational second sub- protocol
Number of newly PCR-confirmed asymptomatic SARS-CoV-2 infection in the observational second sub- protocol | 8 weeks (¨+/- 2 weeks) after 3. vaccination
  Number of newly PCR-confirmed asymptomatic SARS-CoV-2 infection in the observational second sub- protocol

OTHER OUTCOMES:
Safety Outcome: number of local symptoms | during the first 7 days after vaccination
  Any local symptom (redness or swelling or prolonged pain at injection side) limiting continuation of normal daily activities
Safety Outcome: number of systemic symptoms | during the first 7 days after vaccination
  Any systemic symptom (fever, generalized muscle or joint pain) limiting continuation of normal daily activities
Safety Outcome: number of vaccine related symptoms | during the first 7 days after vaccination
  Any vaccine related symptom leading to contacting a physician
Number of participants with newly PCR-confirmed asymptomatic Covid-19 infection (clinical effectiveness endpoint according to FDA recommendations for phase III Covid-19 vaccine licensing trials) | at any time points within 48 weeks follow-up
  Number of participants with newly PCR-confirmed asymptomatic Covid-19 infection (identified by the presence of anti-SARS-CoV-2 nucleocapsid antibodies, or SARS-CoV-" PCR or rapid antigen test) and no related symptoms [(i.e. fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose nausea or vomiting, and diarrhea])
Newly PCR-confirmed symptomatic Covid-19 infection (clinical effectiveness endpoint according to FDA recommendations for phase III Covid-19 vaccine licensing trials) | at any time points within 48 week follow-up
  Newly PCR-confirmed symptomatic Covid-19 infection with at least one of the following symptoms (i.e. fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose nausea or vomiting, and diarrhea)
Number of participants with severe COVID-19 infection (clinical effectiveness endpoint according to FDA recommendations for phase III Covid-19 vaccine licensing trials) | at any time points within 48 week follow-up
  Number of participants with severe COVID-19 infection with respiratory failure, evidence of shock (as diagnosed by a treating physician), clinically significant acute renal, hepatic, or neurologic dysfunction; admission to an intensive care unit; or death
Covid-19 burden of diseases (BOD) (clinical effectiveness endpoint according to FDA recommendations for phase III Covid-19 vaccine licensing trials) | within 48 week follow-up
  Covid-19 burden of diseases (BOD), a composite of the above endpoints. The BOD will be scored as by using 0 for no COVID-19, 1 for non-severe COVID-19, and 2 for severe COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Heiner C. Bucher, Prof. Dr. med., Principal Investigator — Basel Institute for Clinical Epidemiology & Biostatistics, University Hospital Basel
Locations (4):
- Switzerland (4):
  - University Hospital Basel, Basel
  - University Hospital Bern, Bern
  - University Hospital Lausanne CHUV, Lausanne
  - University Hospital Zurich, Zurich

REFERENCES:
- [Result] Speich B, Chammartin F, Abela IA, Amico P, Stoeckle MP, Eichenberger AL, Hasse B, Braun DL, Schuurmans MM, Muller TF, Tamm M, Audige A, Mueller NJ, Rauch A, Gunthard HF, Koller MT, Trkola A, Briel M, Kusejko K, Bucher HC; Swiss HIV Cohort Study and the Swiss Transplant Cohort Study. Antibody Response in Immunocompromised Patients After the Administration of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Vaccine BNT162b2 or mRNA-1273: A Randomized Controlled Trial. Clin Infect Dis. 2022 Aug 24;75(1):e585-e593. doi: 10.1093/cid/ciac169. PMID 35234868
- [Result] Kusejko K, Chammartin F, Smith D, Odermatt M, Schuhmacher J, Koller M, Gunthard HF, Briel M, Bucher HC, Speich B; Swiss HIV Cohort Study; Swiss Transplant Cohort Study. Developing and testing a Corona VaccinE tRiAL pLatform (COVERALL) to study Covid-19 vaccine response in immunocompromised patients. BMC Infect Dis. 2022 Jul 28;22(1):654. doi: 10.1186/s12879-022-07621-x. PMID 35902817
- [Derived] Amstutz A, Chammartin F, Audige A, Eichenberger AL, Braun DL, Amico P, Stoeckle MP, Hasse B, Papadimitriou-Olivgeris M, Manuel O, Bongard C, Schuurmans MM, Hage R, Damm D, Tamm M, Mueller NJ, Rauch A, Gunthard HF, Koller MT, Schonenberger CM, Griessbach A, Labhardt ND, Kouyos RD, Trkola A, Kusejko K, Bucher HC, Abela IA, Briel M, Speich B; Swiss HIV Cohort Study; Swiss Transplant Cohort. Antibody and T-Cell Response to Bivalent Booster SARS-CoV-2 Vaccines in People With Compromised Immune Function: COVERALL-3 Study. J Infect Dis. 2024 Oct 16;230(4):e847-e859. doi: 10.1093/infdis/jiae291. PMID 38848312
- [Derived] Griessbach A, Chammartin F, Abela IA, Amico P, Stoeckle MP, Eichenberger AL, Hasse B, Braun DL, Schuurmans MM, Muller TF, Tamm M, Audige A, Mueller NJ, Rauch A, Gunthard HF, Koller MT, Trkola A, Epp S, Amstutz A, Schonenberger CM, Taji Heravi A, Papadimitriou-Olivgeris M, Casutt A, Manuel O, Kusejko K, Bucher HC, Briel M, Speich B; Swiss HIV Cohort Study and the Swiss Transplant Cohort Study. Antibody Response After the Third SARS-CoV-2 Vaccine in Solid Organ Transplant Recipients and People Living With HIV (COVERALL-2). Open Forum Infect Dis. 2023 Nov 3;10(11):ofad536. doi: 10.1093/ofid/ofad536. eCollection 2023 Nov. PMID 38023564
- [Derived] Chammartin F, Griessbach A, Kusejko K, Audige A, Epp S, Stoeckle MP, Eichenberger AL, Amstutz A, Schoenenberger CM, Hasse B, Braun DL, Rauch A, Trkola A, Briel M, Bucher HC, Gunthard HF, Speich B, Abela IA; Swiss HIV Cohort Study. Bridging the gap: identifying factors impacting mRNA severe acute respiratory syndrome coronavirus 2 vaccine booster response in people with HIV-1. AIDS. 2024 Feb 1;38(2):217-222. doi: 10.1097/QAD.0000000000003751. Epub 2023 Oct 11. PMID 37830908
- [Derived] Chammartin F, Kusejko K, Pasin C, Trkola A, Briel M, Amico P, Stoekle MP, Eichenberger AL, Hasse B, Braun DL, Schuurmans MM, Muller TF, Tamm M, Mueller NJ, Rauch A, Koller MT, Gunthard HF, Bucher HC, Speich B, Abela IA; and the Swiss HIV Cohort Study. Determinants of antibody response to severe acute respiratory syndrome coronavirus 2 mRNA vaccines in people with HIV. AIDS. 2022 Aug 1;36(10):1465-1468. doi: 10.1097/QAD.0000000000003246. Epub 2022 Jul 9. PMID 35876706
- [Derived] Speich B, Chammartin F, Smith D, Stoeckle MP, Amico P, Eichenberger AL, Hasse B, Schuurmans MM, Muller T, Tamm M, Dickenmann M, Abela IA, Trkola A, Hirsch HH, Manuel O, Cavassini M, Hemkens LG, Briel M, Mueller NJ, Rauch A, Gunthard HF, Koller MT, Bucher HC, Kusejko K; study groups from the Swiss HIV Cohort Study and the Swiss Transplant Cohort Study. A trial platform to assess approved SARS-CoV-2 vaccines in immunocompromised patients: first sub-protocol for a pilot trial comparing the mRNA vaccines Comirnaty(R) and COVID-19 mRNA Vaccine Moderna(R). Trials. 2021 Oct 21;22(1):724. doi: 10.1186/s13063-021-05664-0. PMID 34674742

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Sub-Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT04805125/Prot_SAP_000.pdf
  • Study Protocol: Master-Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT04805125/Prot_001.pdf
  • Study Protocol: Second Sub-Protocol (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT04805125/Prot_002.pdf
  • Study Protocol: Third Sub-Protocol (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT04805125/Prot_003.pdf